CLINICAL TRIAL: NCT02369822
Title: Trial of Vitamin C as Add on Therapy for Children With Idiopathic Epilepsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shaymaa Maher Deifalla, Lecturer of Pediatrics, Faculty of Medicine, Ain Shams University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin C, Children, Epilepsy
Record Dates: First submitted 2015-02-11; First posted 2015-02-24 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Idiopathic Epilepsy
Keywords: Vitamin C; convulsions status; EEG; children
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin C supplemented (Experimental): patients with refractory idiopathic epilepsy will receive vitamin C supplement according to age for 1 month
  Interventions: Dietary Supplement: Vitamin C
- None supplemented (No Intervention): followed up for 1 month

INTERVENTIONS:
Dietary Supplement: Vitamin C — those who are 2-3 years will receive 400 mg/day, 4-8 years will receive 500 mg/day, those who are 9-13 years will receive 1000 mg/day, and from 14-16 years will receive 1500 mg/day
  Arms: Vitamin C supplemented

SUMMARY:
There are no solid treatment guidelines for idiopathic intractable epilepsy in children. The investigators propose that vitamin C being an antioxidant will improve seizure frequency and EEG in children with idiopathic intractable epilepsy.

DETAILED DESCRIPTION:
Is vitamin C; being an antioxidant based on the hypothesis of oxidative stress as a provocation factor for idiopathic epilepsy low in those with idiopathic epilepsy, and is it lower in those with refractory than those with newly diagnosed? Will vitamin C supplementation for 1 month be efficient to raise the vitamin C level and will it improve seizures and EEG findings in those with idiopathic epilepsy?

ELIGIBILITY:
Inclusion Criteria:

* Normal neuroimaging

Exclusion Criteria:

* Developmental delay.
* Suspected metabolic problems.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-09 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Seizure severity and frequency, EEG findings | up to 30 days
  Seizure severity based on the Chalfont seizre severity scale and daily seizure frequency will be measured before and 30 days after vitamin C supplementation in children with intractable idiopathic epilepsy

SECONDARY OUTCOMES:
vitamin C level in children with epilepsy | 6 months
  children with epilepsy will be recruited over a period of 6 months and we will measure vitamin C level in their blood

CONTACTS AND LOCATIONS:
Overall Officials: Iman A Elagouza, A Professor, Study Director — Faculty of Medicine, Ain Shams University
Locations (1):
- Shaymaa Maher Deifalla, Cairo, Nasr City, Egypt